CLINICAL TRIAL: NCT00488397
Title: Tigecycline In-Vitro Surveillance Study In Taiwan
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Other Study IDs: 3074A1-102091; B1811055 (Other: Pfizer)
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2011-03

CONDITIONS: Community Acquired Infections
Keywords: Tygacil; microdilution method; Tigecycline; In-Vitro
MeSH Terms: conditions — Community-Acquired Infections | interventions — In Vitro Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Other: In-vitro testing

INTERVENTIONS:
Other: In-vitro testing — This is an in-vitro study thus only one group in the study and there is no intervention treatment nor procedure involved in this study.

SUMMARY:
In-vitro surveillance study of tigecycline (Tygacil) in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Clinically relevant causative isolate (no duplicates) - The isolate must meet the laboratory criteria of "significant pathogen" and be considered the "probable causative agent" of a hospital or community acquired infection.
* Sources - All body sites are acceptable clinical sources for isolates to be included in this study (Intra-abdominal infection, tracheal secretion/bronchoalveolar lavage, blood culture, wound smear). However, no more than 10 % of all isolates can come from urine cultures.
* Within study group - Only isolates defined by the protocol are to be included.

Exclusion Criteria:

* Limited isolates from sources - No more than 10 % of all isolates from this study will be derived from urine cultures.
* No banked or stored isolates.
* No duplicate isolates - Only one isolate per patient is permitted.
* Outside study group - Any isolate other than those defined by protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: hospital or community acquired infection
Sampling Method: Non-Probability Sample
Enrollment: 7902 (Actual)
Dates: Start 2006-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Prior to 2009: Susceptibility data of minimum inhibitory concentration (MIC), MIC50, MIC90by pathogen, tested by E-test. | in vitro study therefore not applicable
Post-2009: Susceptibility data of MIC, MIC50, MIC90 by pathogen, tested by micro-dilution method | in vitro study therefore not applicable

SECONDARY OUTCOMES:
Prior to 2009: 1. Susceptibility data of minimum inhibitory concentration (MIC), MIC50, MIC90 by pathogen, tested by micro-dilution method 2. Susceptibility data of inhibition zone diameter(mm) by pathogen, tested by paper disc. | in vitro study therefore not applicable
Post-2009: Susceptibility data of inhibition zone diameter (mm) by pathogen, tested by paper disc. | in vitro study therefore not applicable

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Taipei, Taiwan, China

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3074A1-102091&StudyName=Tigecycline%20In-Vitro%20Surveillance%20Study%20In%20Taiwan